CLINICAL TRIAL: NCT03423602
Title: Clinical Investigation Plan (CIP) for Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER IV Study
Brief Title: Safety and Performance Study of Large Hole Vascular Closure Device FIV
Acronym: Frontier-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P528-00
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Percutaneous CFA Arteriotomy Closure
Keywords: Percutaneous vascular closure device; Large hole closure device; Arteriotomy closure; Vascular closure device

STUDY DESIGN:
Intervention Model Description: prospective, multi-centred, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational device (Experimental): To confirm safety and performance of the PerQseal® Closure Device (DP2-FA1-4) and PerQseal® Introducers (DP2-FA1-5 and DP2-FA1-6) to percutaneously close femoral artery punctures and to induce arterial haemostasis in patients undergoing endovascular procedures requiring an arteriotomy created by 12 to 20 F sheaths.
  Interventions: Device: PerQseal®

INTERVENTIONS:
Device: PerQseal® — Large hole closure system
  Other Names: DP2-FA1-4 DP2-FA1-5 DP2-FA1-6

SUMMARY:
The purpose of this Clinical Investigation Plan (CIP) is to:

1. Confirm the safety and performance of the PerQseal® large hole closure system.
2. To expand its indications of use to include common femoral arteriotomies created with 12 to 20 F sheaths in patients undergoing endovascular procedures.

DETAILED DESCRIPTION:
This study will be a prospective, multi-centred, non-randomized study to investigate the safety and performance of the PerQseal® in 75 patients in approximately 10 European investigational sites.

The study shall not be blinded prior to, during or post the procedure. All patients undergoing an endovascular procedure requiring an arteriotomy created by 12 to 20 F sheaths, via the common femoral artery will be screened against the inclusion/exclusion criteria. If the patient meets the requirements of the clinical investigation, they shall be invited to participate, provide informed consent and shall subsequently be assigned a subject number.

All subjects shall have an immediately post procedure, ~24 hour, 1 and 3 month follow-up assessment. Safety data from the follow-ups will be assessed by the Data Safety Monitoring Committee on a continuous basis.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
* Clinically indicated for an endovascular procedure using a common femoral arteriotomy created by a 12 - 20 F sheath.

Exclusion Criteria:

* Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than six months.
* Evidence of systemic bacterial or cutaneous infection, including groin infection.
* Known bleeding diathesis, definite or potential coagulopathy, platelet count < 100,000/μl or patients on long term anticoagulants with an INR greater than 1.2 at time of procedure or known type II heparin-induced thrombocytopenia.
* Severe; claudication or peripheral vascular disease (e.g. Rutherford category 3 or greater or ABI < 0.5), documented untreated iliac artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of ipsilateral limb.
* Known allergy to any of the materials used in the PerQseal®.
* Subject has undergone a percutaneous procedure using a non-absorbable vascular closure device (excluding suture mediated) for haemostasis in the ipsilateral target leg.
* Patients that have undergone a percutaneous procedure in the ipsilateral leg, within the previous 30 days.
* Patients that have undergone a percutaneous procedure using an absorbable intravascular closure device for haemostasis, in the ipsilateral leg, within the previous 90 days.
* Evidence of arterial diameter stenosis > 20% or anterior or circumferential calcification within 20 mm proximal or distal to target arteriotomy site based on pre-procedure CT angiography.
* Females who are pregnant or lactating or in fertile period not taking adequate contraceptives. A pregnancy test may be performed.
* Patients that have a lower extremity amputation from the ipsilateral or contralateral limb.
* Arterial access other than common femoral artery obtained for ipsilateral target leg.
* Subject has a tissue tract expected to be greater than 10 cm.
* Use of thrombolytic agents within 24 hours prior to or during the endovascular procedure which causes fibrinogen < 100 mg/dl.
* Significant blood loss/transfusion (defined as requiring transfusion of 4 or more units of blood products) during index procedure or within 30 days prior to index procedure.
* Activated clotting time (ACT) > 350 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 350 seconds for more than 24 hours after index procedure.
* Target puncture site is located in a vascular graft.
* Target arteriotomy in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 10 mm proximal of the bifurcation of the Superficial Femoral /Profunda Femoris artery.
* PerQseal® Introducer-sheath to ipsilateral femoral artery diameter ratio is greater than or equal to 1.05.
* Subjects with an acute haematoma of any size, arteriovenous fistula or pseudoaneurysm at the target access site; or angiographic evidence of arterial laceration or dissection within the external iliac or femoral artery before the use of the PerQseal® closure device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Arne Schwindt, Principal Investigator — St Fraziskus Hospital, Muenster, Germany; Dr Christoph Naber, Principal Investigator — Contilia Heart and Vascular centre, Essen, Germany
Locations (11):
- Germany (9):
  - Kerckhoff Klinik, Bad Nauheim, Bad Nauheim, Hesse
  - CardioVasculäres Centrum, Frankfurt am Main, Hesse
  - Uniklinik Köln, Herzzentrum, Cologne, North Rhine-Westphalia
  - Contilia Heart and Vascular centre, Essen, North Rhine-Westphalia
  - St Franziskus Hospital, Münster, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Medical Faculty of the University of Leipzig, Leipzig, Saxony
  - The Charité - Universitätsmedizin, Mitte, State of Berlin
  - Asklepios Klinik St. Georg Medizinische Abteilung, Hamburg
- Ireland (2):
  - Blackrock Clinic, Blackrock, Dublin
  - St James Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from each of the participating centres undergoing an endovascular interventional procedure requiring a percutaneous common femoral arterial access using sheath sizes in the range of 12 to 20 F were screened against the inclusion/exclusion criteria for eligibility. If a patient met the requirements of the clinical investigation, they were invited to participate, given patient information relative to the study and if willing to participate were asked to sign informed consent.
Pre-assignment Details: Subjects with bilateral percutaneous access in both common femoral arteries, where both arteries met all eligibility criteria, were closed bilaterally with the Investigational device, at the discretion of the investigator. If a test device was used on both ipsilateral and contralateral femoral arteries, then each closure (i.e. each limb) was treated as an independent closure.
Units Other Than Participants: Limbs
Period: Overall Study
Arm/Group | Investigational Device
Started | 75; 84 Limbs
Discharge | 70; 77 Limbs (One subject died prior to discharge: due to cerebral infarction following cardiac arrest, not related to the study device. Four subjects were excluded from the study with no further follow-up due to not being implanted with a study device.)
1-month Follow-up | 66; 71 Limbs (Two subjects voluntarily withdrew their consent to remain in the study. One subject was excluded from the study post discharge examination due to unrelated groin surgery. One subject was not followed-up at 1-month due to unrelated gastrointestinal complications (and subsequently withdrew from the study prior to 3-month follow-up); Three subjects missed their 1-month follow-up, however remained in the study and attended their 3-month follow-up assessment.)
3-month Follow-up | 63; 72 Limbs (Two subjects voluntarily withdrew their consent to remain in the study. One subject was lost to follow-up)
Completed | 63; 72 Limbs
Not Completed | 12; 12 Limbs
Not completed — Death | 1
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Device
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Procedure
  years | 78.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ireland | 5
  Germany | 70
Primary Procedure type [Count of Participants; unit: Participants] — Patient cohorts included within the study are: Endovascular Aortic Aneurysm Repair (EVAR), Thoracic Endovascular Aortic Aneurysm Repair (TEVAR), Transcatheter Aortic Valve Repair (TAVR)
  Participants
    TAVR | 41
    EVAR | 30
    TEVAR | 4
Height [Mean (Standard Deviation); unit: cm] | 170.1 (9.4)
Weight [Mean (Standard Deviation); unit: kg] | 80.8 (15.3)
Co-morbidity [Count of Participants; unit: Participants]
  Hypertention | 65
  Diabetes | 22
  Severe acute non-cardiac systemic disease, autoimmune disease or terminal illness | 0
  Clinically significant peripheral vascular disease | 2
  Bleeding diatheses | 2
  Previous peripheral vascular surgery involving the aorta or lower extremities | 4
  Claudication | 1

OUTCOME MEASURES:

1. Primary Outcome: Major Vascular Complications [Safety]
Description: Rate of major vascular access site complications related to the PerQseal® closure device (as defined by VARC-2)
Time Frame: up to 1 month post implantation
Population: All enrolled subjects with any major device related event. Includes all subjects through the last assessment prior to or at 1-month post implantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device
Number analyzed (Participants) | 75
Participants | 0
Statistical Analysis 1: Comparison: Investigational Device; The test for non-inferiority for safety was based on a one-sided test (at the 0.025 significance level) for a binomial proportion with hypotheses: H0s: Psafety ≥ NLs versus H1s: Psafety < NLs Where: Psafety is the actual proportion of device related major vascular access site complications within the study population; and NLs is the non-inferiority limit for proportion of expected major vascular access site complications associated with cut-down and suture closure; Test type: Non-Inferiority — Based on a Meta-Analysis of a focused systematic literature review from a comparable patient population, the estimated major vascular access site complication rate or PGsafety for the conservative Random Effect Model is 0.125 with a 95% Confidence Interval of 0.09 to 0.17. Given that the upper bound was 0.17 this justified the use of 0.13 as a valid PGsafety plus a non-inferiority margin of 0.04 yielding an overall non-inferiority limit (NLs) of 0.17 for Safety. Study power is greater than 90%; p < .0001, Wilson's exact test; All 75 enrolled subjects, regardless of their enrolment status at 1-month post implantation, including all reported safety data where included; Wilson's exact test = 0.0487, 95% CI 1-sided [upper limit 0.0487]

2. Secondary Outcome: Minor Vascular Complications [Safety]
Description: Rate of minor vascular access site complications directly related to the PerQseal® closure device (as defined by VARC-2)
Time Frame: up to 1 month from implantation
Population: All subjects with any minor device related event. Includes all subjects through the last assessment prior to or at 1-months
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device
Number analyzed (Participants) | 75
Participants
  All enrolled subjects | 5
  Subjects still enrolled at 1-month with follow-up: number analyzed (Participants) | 63
  Subjects still enrolled at 1-month with follow-up | 3

3. Secondary Outcome: Study Device Technical Success Rate [Performance]
Description: Percentage of closures (Limbs) with Technical Success, for the PerQseal® closure device, not requiring alternative therapy to achieve haemostasis
Time Frame: within 24 hours
Population: Technical success analysis included all closures that received the investigational device (79)
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Investigational Device
Number analyzed (Participants) | 75
Number analyzed (Limbs) | 79
Limbs | 75

ADVERSE EVENTS:
Time Frame: From Subject enrolment to study exit which was 3-months ± 1-month
Description: Adverse Event definitions where those given in ISO 14155:2011. All adverse events were reported via the eCRF, whether or not they were related to the use of the test device or access closure procedure. All complications, SAEs, SADEs and USADEs were reviewed on a continuous basis by an independent Data Safety Monitoring Committee. All access site related complications were reviewed and adjudicated by an independent Clinical Events Committee. All safety data was 100% SDV during monitoring.
Arm/Group | Investigational Device
All-Cause Mortality (participants affected / at risk) | 1/75
Serious Adverse Events (participants affected / at risk) | 21/75
Other Adverse Events (participants affected / at risk) | 5/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=75)
Cardiac decompensation (Cardiac disorders) | 4 (4)
Lymphocele (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated to investigational device
Access site haematoma (Vascular disorders) | 3 (3) — Two related to investigational closure device
Aneurysm (Vascular disorders) | 2 (2) — Not access site or target vessel
Arrhythmia - AV Block (Cardiac disorders) | 3 (3)
Arteriovenous fistula - access site (Vascular disorders) | 1 (1) — Not related to investigational closure device
Cardiac tamponade (Cardiac disorders) | 1 (1)
Dissection (Vascular disorders) | 1 (1) — Not access site or target vessel
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) — Not access site or target vessel
Hypertension (Vascular disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Graft occlusion (Vascular disorders) | 1 (1) — Not access site or target vessel
Infection (Infections and infestations) | 1 (1) — Not related to access closure. Related to post surgical intervention
Renal failure (Renal and urinary disorders) | 1 (1)
Septicaemia (Blood and lymphatic system disorders) | 2 (2)
Spinal anterior syndrome (Nervous system disorders) | 1 (1)
Stroke - ischemic (Vascular disorders) | 1 (1)
Urinary infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=75)
Haematoma (Vascular disorders) | 3 (3) — Minor access site complication. Relationship to device: 1 x Probable, 2 x Possible
Pseudoaneurysm (Vascular disorders) | 2 (2) — Minor access site complication. Relationship to device: 1 x Causal, 1 x Probable

LIMITATIONS AND CAVEATS:
Study was a single-arm study precluding any direct comparison with other VCDs. Patient population was selected based on inclusion/exclusion including a restriction of the Sheath to Femoral Artery Ratio greater than 1.05 and anterior or circumferential calcification at or near the access site. There are a relatively small number of subjects with a BMI greater than 30 in the study population. There was a relatively small number of subjects in the study with a primary sheath size greater than 19 F.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03423602/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03423602/SAP_001.pdf